CLINICAL TRIAL: NCT03979352
Title: Effect of SGLT2 Inhibition on Improving the Glycemic Performance of the Single Hormone Artificial Pancreas Configuration in Type 1 Diabetes in the Outpatient Setting - A Randomized Placebo Controlled Cross-Over Multicentre Clinical Trial
Brief Title: Effect of SGLT2i in Conjunction With the Artificial Pancreas on Improving the Glycemia in T1DM in the Outpatient Setting
Acronym: CLASS17
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Collaborators: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CLASS 17
Record Dates: First submitted 2019-04-13; First posted 2019-06-07 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2019-11

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Empagliflozin; Artificial Pancreas; SGLT2 inhibitor; insulin pump; closed loop
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — empagliflozin; Pancreas, Artificial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Empagliflozin arm (Active Comparator): Participant will be treated by empagliflozin for 8 weeks. During these 8 weeks he will use artificial pancreas to deliver the insulin for 4 weeks and conventional pump therapy for remaining 4 weeks, in a random order.
  After finishing the entire arm intervention participant will undergo 7 day of washout and enters the placebo arm.
  Participant and research staff is blinded to arm assignment.
  Interventions: Drug: empagliflozin; Device: artificial pancreas
- Placebo arm (Placebo Comparator): Participant will take placebo for 8 weeks. During these 8 weeks he will use artificial pancreas to deliver the insulin for 4 weeks and conventional pump therapy for remaining 4 weeks, in a random order.
  After finishing the entire arm intervention participant will undergo 7 day of washout and enters the empagliflozin arm.
  Participant and research staff is blinded to arm assignment.
  Interventions: Device: artificial pancreas

INTERVENTIONS:
Drug: empagliflozin — Treatment with empagliflozin 25mg orally once a day
  Arms: Empagliflozin arm
Device: artificial pancreas — Insulin delivery via a closed loop single-hormone artificial pancreas system.

SUMMARY:
The most advanced configurations of the Artificial Pancreas (AP) have not yet been demonstrated to sufficiently maximize time in target glycemia. One limitation is the challenge of postprandial glycemic control, which currently requires ongoing patient engagement for accurate and detailed bolus dose estimation for meals. Sodium Glucose Linked Transporter 2 Inhibition (SGLT2i) provides an additional mechanism to attenuate post-prandial glycemic excursion, and may represent a strategy that could further alleviate carbohydrate counting burden and improve the performance of AP configurations. This trial aims to compare - using a randomized, masked placebo-controlled, crossover, multicenter design - the efficacy of the SGLT2i empagliflozin 25 mg oral per day each in the setting of single-hormone automated AP and conventional insulin pump therapy on the proportion of time spent in target and in hypoglycemia each during a 4-week day-and-night period. The pilot trial aims to enroll 28 adult patients with type 1 diabetes (T1D) across 2 research sites (one in Toronto and one in Montreal) and includes a 2- week therapy optimization run-in period, 4-weeks for each of the two AP intervention arms, and a 1- week washout in between the pharmacological intervention sequences. Glucose levels will be measured by continuous glucose monitoring (G5, Dexcom Inc.). Insulin will be infused using a subcutaneous infusion pump (t-slim, Tandem Diabetes Care) and communication between pumps and the algorithm will be implemented using Android Smartphone devices and Bluetooth technology communication.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated written informed consent by the date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation.
2. Males and females ≥ 18 years of age.
3. Clinical diagnosis of T1D for at least one year. The diagnosis of T1D is based on the investigator's clinical judgment; C peptide level and antibody determinations are not planned.
4. Insulin pump therapy use for at least 3 months.
5. HbA1c ≤ 10%.
6. eGFR ≥ 60 mL/min/1.73 m² as calculated by the CKD-EPI formula.
7. Women of child-bearing potential must be ready and able to use highly effective methods of birth control that result in a low failure rate of less than 1% per year when used consistently and correctly.

Exclusion Criteria:

1. Clinically significant nephropathy, neuropathy or retinopathy as judged by the investigator.
2. Recent (< 6 months) acute macrovascular event e.g. acute coronary syndrome or cardiac surgery.
3. Renal insufficiency (characterized at eGFR below 60 mmol/l at the beginning of the trial)
4. History of pheochromocytoma or insulinoma
5. Beta-blockers at high dose (interference with glucose management).
6. Chronic acetaminophen treatment (can interfere with glucose sensor measurements).
7. Warfarin chronic treatment if INR monitoring cannot be evaluated (can increase the risk of bleeding).
8. Current use of other non-insulin adjunct anti-hyperglycemic drug or use within 30 days prior to screening.
9. Use of loop diuretics (e.g. furosemide, due to possible interference with study drug mechanism of action).
10. Ongoing or planned pregnancy or breastfeeding.
11. Severe hypoglycemic episode within one month prior to Visit 1.
12. Diabetic ketoacidosis in the last 3 months prior to Visit 1.
13. Current use of glucocorticoid medication except low stable dose and inhaled steroids (can interfere with glucose sensor measurements).
14. Known or suspected allergy to the trial products.
15. Other serious medical illness likely to interfere with study participation or with the ability to complete the trial by the judgment of the investigator.
16. Anticipating a significant change in exercise regimen between initiation of two intervention blocks (i.e. starting or stopping an organized sport).
17. Recent history of genital or urinary infection (<1 month prior to Visit 1) or history of recurrent urinary tract infections.
18. Difficulty in using the artificial pancreas system following training.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in sensor glucose target range defined as between 3.9 and 7.8 mmol/L compared between 4- weeks AP on empagliflozin and 4-weeks AP with placebo | 20 weeks
  Percentage of time spent in sensor glucose target range defined as between 3.9 and 7.8 mmol/L compared between 4- weeks AP on empagliflozin and 4-weeks AP with placebo.
Percentage of time spent in sensor glucose target range defined as between 3.9 and 7.8 mmol/L compared between 4- weeks conventional pump therapy on empagliflozin and 4- weeks conventional pump therapy with placebo | 20 weeks
  Percentage of time spent in sensor glucose target range defined as between 3.9 and 7.8 mmol/L compared between 4- weeks conventional pump therapy on empagliflozin and 4- weeks conventional pump therapy with placebo.
Percentage of time spent in sensor glucose target range defined as between 3.9 and 7.8 mmol/L on 4- weeks automated AP on empagliflozin when compared to 4-weeks conventional pump therapy on empagliflozin | 20 weeks
  Percentage of time spent in sensor glucose target range defined as between 3.9 and 7.8 mmol/L on 4- weeks automated AP on empagliflozin when compared to 4-weeks conventional pump therapy on empagliflozin.
Percentage of time spent in sensor glucose target range defined as between 3.9 and 7.8 mmol/L on 4- weeks automated AP on empagliflozin when compared to 4-weeks conventional pump therapy with placebo | 20 weeks
  Percentage of time spent in sensor glucose target range defined as between 3.9 and 7.8 mmol/L on 4- weeks automated AP on empagliflozin when compared to 4-weeks conventional pump therapy with placebo.

SECONDARY OUTCOMES:
Percentage of time spent in sensor glucose target range defined as between 3.9 and 10.0 mmol/L compared between 4- weeks conventional pump therapy on empagliflozin and 4-weeks AP on empagliflozin | 20 weeks
  Percentage of time spent in sensor glucose target range defined as between 3.9 and 10.0 mmol/L compared between 4- weeks conventional pump therapy on empagliflozin and 4-weeks AP on empagliflozin
Percentage of time spent in sensor glucose target range defined as between 3.9 and 10.0 mmol/L compared between 4- weeks AP on empagliflozin and 4- weeks AP with placebo | 20 weeks
  Percentage of time spent in sensor glucose target range defined as between 3.9 and 10.0 mmol/L compared between 4- weeks AP on empagliflozin and 4- weeks AP with placebo.
Hypoglycemia: Percentage of time with glucose <3.9 mmol/L applied to each of the primary and secondary outcome comparator groups | 20 weeks
  Hypoglycemia: Percentage of time with glucose <3.9 mmol/L applied to each of the primary and secondary outcome comparator groups.
Percentage of time spent in hypoglycemia, euglycemia and hyperglycemia | 20 weeks
  Percentage of time spent in the different glucose sensor levels characterized by amount spent between 3.9 and 10.0 mmol/L, 3.9 and 7.8 mmol/L, above 10.0 mmol/L, above 13.9 mmol/L, above 16.7 mmol/l, below 3.9 mmol/L, below 3.3 mmol/L, below 2.8 mmol/L
Absolute number of hypoglycemia events I. | 20 weeks
  Number of hypoglycemic events (> 20 minutes) below 3.3 mmol/L based on sensor glucose levels
Absolute number of hypoglycemia events II. | 20 weeks
  Number of symptomatic hypoglycemic events < 3.9 mmol/l or below 3.3 mmol/l without symptoms
Absolute number of hypoglycemia events III. | 20 weeks
  Number of treated hypoglycemic events
Statistical characteristics of glucose profile I. | 20 weeks
  Area under the curve of hypoglycemic glucose values (below 3.9 mmol/L, 3.3 mmol/L and 2.8 mmol/L)
Statistical characteristics of glucose profile II. | 20 weeks
  Standard deviation of glucose levels
Amount of total insulin delivery during interventions | 20 weeks
  Total insulin delivery measured by mean of units per day
Change in HbA1c | 20 weeks
  Change in HbA1c from baseline to after the first intervention and from the end of the first intervention to the end of the treatment period.
Mean fasting capillary ketone levels | 20 weeks
  Mean fasting capillary ketone levels.
Number of episodes of diabetic ketoacidosis | 20 weeks
  Number of episodes of diabetic ketoacidosis
Number of technical adverse events | 20 weeks
  Number of events when algorithm crashes or needs to be overridden for safety reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Perkins, MD, Principal Investigator — Samuel Lunenfeld Research Institute
Locations (2):
- Canada (2):
  - Sinai Health System, Toronto, Ontario
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No